CLINICAL TRIAL: NCT07335510
Title: Impact of Barostimulation in Cardiac Hemodynamics and Clinical Outcomes Through Use of the Barostim™ CVRx Device
Brief Title: Impact of Barostimulation on Hemodynamics in Adults With Heart Failure
Acronym: BREATHE-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: CVRx, Inc. (Industry)
Responsible Party: Principal Investigator, Nir Uriel, Professor of Cardiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV9622
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: HFrEF - Heart Failure With Reduced Ejection Fraction
Keywords: Baroreflex activation therapy; Exercise hemodynamics; Barostim; Cardiopulmonary exercise testing; Neuromodulation; Functional capacity; Heart failure with reduced ejection fraction

STUDY DESIGN:
Intervention Model Description: This is a single-group, self-controlled study in which all enrolled participants receive the same intervention. Outcomes are evaluated within participants using pre- and post-implantation assessments following Barostim device implantation and titration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Barostim™ Therapy (Experimental): Participants will undergo implantation of the Barostim™ system, followed by device programming and titration according to standard clinical practice for up to three months after implantation.
  Interventions: Device: Baroreflex Activation Therapy

INTERVENTIONS:
Device: Baroreflex Activation Therapy — Barostim™ device (CVRx Inc.), a commercially available, FDA-approved device for autonomic modulation in HFrEF. The device system includes an implantable pulse generator, carotid sinus lead, and programmer system. No investigational modifications will be made. The device will be implanted per standard labeling and programming guidelines, and therapy titration will follow manufacturer recommendations.

SUMMARY:
This study evaluates the effects of the implantation and adjustment of the CVRx Barostim device in adult patients with heart failure with reduced ejection fraction who are receiving maximally tolerated doses of guideline directed medical and device therapies. The study aims to assess how therapy using this device affects heart function, symptoms, and exercise capacity, with particular focus on how the device affects blood flow and heart pressures during exercise. Information from this study may help inform patient selection and device management in patients with heart failure.

DETAILED DESCRIPTION:
Heart failure with reduced ejection fraction (HFrEF) remains a major public health concern, associated with high rates of morbidity, hospitalizations, and mortality. Despite advances in medication, as well as device therapies such as implantable devices, a significant proportion of patients continue to experience debilitating symptoms, exercise intolerance, and reduced quality of life.

An important feature of HFrEF is autonomic imbalance, which contributes to disease progression and adverse outcomes. While current therapies indirectly try to affect this imbalance, the Barostim™ device (CVRx) is the first to specifically target the autonomic nervous system in this population. This device offers a novel mechanistic approach by directly stimulating the carotid baroreceptors to reduce sympathetic activity and restore autonomic balance. This prospective multicenter study aims to evaluate the effects of the Barostim device on invasive hemodynamics through right heart catheterization (RHC), exercise capacity, and tolerance to medical therapy in HFrEF patients who remain symptomatic despite maximal guideline-directed medical therapy (GDMT). The study seeks to address key knowledge gaps in the mechanistic and clinical response to baroreflex activation therapy (BAT) and inform future integration of this therapy into standard heart failure care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure with reduced ejection fraction (defined as ejection fraction ≤ 35% for the purposes of this study) (should be within 12 months of screen)
* Symptoms consistent with one of:

  1. current New York Heart Association (NYHA) Class III or
  2. current NYHA Class II and historical NYHA Class III
* Laboratories with last N-terminal pro-B-type natriuretic peptide (NT-proBNP) < 1600 pg/ml (should be within 3 months of screen)
* Management with maximally-tolerated GDMT medications and devices
* Age >= 18 years

Exclusion Criteria:

* Age < 18 years
* Myocardial infarction (MI), syncope, cerebrovascular accident (CVA), aborted sudden cardiac death (SCD) (and implantable cardioverter defibrillator (ICD) therapy) within 3 months of screening
* Bilateral carotid bifurcations located above the level of the mandible
* Carotid artery stenosis greater than 50% caused by atherosclerosis
* Ulcerative plaques in the carotid artery
* Baroreﬂex failure or autonomic neuropathy
* Symptomatic un-controlled bradyarrhythmias
* Severe chronic lung disease
* Current treatment with inotropes
* Pacemaker or ICD within 3 months of screening
* Cardiac resynchronization therapy (CRT) devices within 6 months of screening or anticipated to be placed in the next 90 days following screening
* Prior surgery, radiation, endovascular stent in the carotid sinus
* History or consideration of solid organ transplantation
* History or consideration of left ventricular assist device (LVAD)
* Life expectancy <1 year from time of screening
* Non-cardiovascular conditions interfering with 6MWT distance assessment
* Inability to fulﬁll protocol requirements
* Known allergy to silicone or titanium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in peak exercise PCWP at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Exercise pulmonary capillary wedge pressure (PCWP) will be measured at peak exercise at approximately six months post-Barostim titration and compared with peak exercise PCWP measured during the pre-implantation phase. Change from baseline will be calculated.

SECONDARY OUTCOMES:
Change in peak exercise load-adjusted PCWP at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Exercise pulmonary capillary wedge pressure (PCWP) will be measured at peak exercise at approximately six months post-Barostim titration and compared with peak exercise PCWP measured during the pre-implantation phase. PCWP measurements will be normalized to maximal exercise load at each time point. Change from baseline will be calculated.
Change in peak exercise output-adjusted PCWP at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Exercise pulmonary capillary wedge pressure (PCWP) will be measured at peak exercise at approximately six months post-Barostim titration and compared with peak exercise PCWP measured during the pre-implantation phase. PCWP measurements will be normalized to cardiac output at each time point. Change from baseline will be calculated.
Change in peak exercise cardiac output at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Exercise cardiac output (CO) will be measured at peak exercise at approximately six months post-Barostim titration and compared with peak exercise CO measured during the pre-implantation phase. Change from baseline will be calculated.
Proportion of participants with significant reduction in PCWP at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Exercise pulmonary capillary wedge pressure (PCWP) will be measured at peak exercise at approximately six months post-Barostim titration and compared with peak exercise PCWP measured during the pre-implantation phase. Patients will be categorized into "responders" who demonstrate either a 10% reduction in PCWP or a 3 mmHg reduction in PCWP or "non-responders" who do not demonstrate at least this degree of percent or absolute change. The proportion of participants that are considered "responders" by this metric will be collected and assessed.
Change in peak exercise mean PA pressures at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Exercise mean pulmonary arterial pressure (PAP) will be measured at peak exercise at approximately six months post-Barostim titration and compared with peak exercise mean PAP measured during the pre-implantation phase. Change from baseline will be calculated.
Change in peak VO2 at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Exercise peak VO2 will be measured via cardiopulmonary exercise testing (CPET) at approximately six months post-Barostim titration and compared with peak VO2 measured via CPET during the pre-implantation phase. Change from baseline will be calculated.
Change in average daily step count | Pre-implantation phase (baseline, 0-2 months) and post-implantation phase monthly (approximately 0-9 months post-implantation).
  Average daily step counts will be measured via study-provided Fitbit Inspire 3 fitness trackers. Absolute change and trends will be assessed from baseline to monthly time points in the post-implantation phase.
Change in average daily step count at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  The most recent 30-day period of daily step counts will be measured via study-provided Fitbit Inspire 3 fitness trackers and evaluated for the average daily step count. This will be assessed at approximately six months post-Barostim titration and compared with the average of the last 30-day period of daily step counts prior to the end of the pre-implantation phase. Change from baseline will be calculated.
Change in highest daily step count at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  The most recent 30-day period of daily step counts will be measured via study-provided Fitbit Inspire 3 fitness trackers and evaluated for the maximum daily step count. This will be assessed at approximately six months post-Barostim titration and compared with the maximum of the last 30-day period of daily step counts prior to the end of the pre-implantation phase. Change from baseline will be calculated.
Change in estimated peak VO2 at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  The most recent Fitbit cardio fitness score (estimated peak VO2) will be measured via study-provided Fitbit Inspire 3 fitness trackers. This will be assessed at approximately six months post-Barostim titration and compared with the most recent Fitbit cardio fitness score prior to the end of the pre-implantation phase. Change from baseline will be calculated.
Change in heart rate variability at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  The most recent 30-day average of heart rate variability will be measured via study-provided Fitbit Inspire 3 fitness trackers. This will be assessed at approximately six months post-Barostim titration and compared with the average of the last 30-day period prior to the end of the pre-implantation phase. Change from baseline will be calculated.
Change in proportion of exercise days per month at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  The most recent 30-day proportion of exercise days will be measured via study-provided Fitbit Inspire 3 fitness trackers. This will be assessed at approximately six months post-Barostim titration and compared with the proportion of exercise days of the last 30-day period prior to the end of the pre-implantation phase. Change from baseline will be calculated.
Change in six-minute walk test at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  A six-minute walk test (6MWT) will be performed, and distances will be measured. This will be assessed at approximately six months post-Barostim titration and compared with the 6MWT performed during the pre-implantation phase. Change from baseline will be calculated.
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ)-12 at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  The KCCQ in its 12-question version will be performed to assess quality of life, and each question has 5-7 Likert-style response options. Responses are grouped according to domain for domain-specific scores. Overall and domain-specific scores are transformed and standardized and final scores are reported from 0-100, where higher scores reflect less functional limitation and better quality of life (better outcome). This will be assessed at approximately six months post-Barostim titration and compared with the KCCQ scores obtained during the pre-implantation phase. Change from baseline will be calculated.
Change in heart failure medication score at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  A heart failure medication score (0-9 points) will be calculated based upon participants' current heart failure medications, with 9 indicating a better outcome. Scored are allocated in the following manner: 2 points for being on a mineralocorticoid receptor antagonist or a sodium-glucose cotransporter 2 inhibitor; 2 points for being on a heart failure-specific beta blocker (carvedilol, metoprolol succinate, or bisoprolol; 2 points for >= 50% max guideline-directed dose, 1 point for <50% dose, 0 points if not); and 3 points for being on a renin-angiotensin-aldosterone system inhibitor (3 points for an angiotensin receptor-neprilysin inhibitor, or 1-2 points for either an angiotensin-converting-enzyme inhibitor or an angiotensin receptor blocker at <50% or >=50% max guideline-directed dose). This will be assessed at approximately six months post-Barostim titration and compared with the medication scores obtained during the pre-implantation phase. Change from baseline will be calculated.
Change in N-terminal prohormone of brain natriuretic peptide at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Participants' levels of N-terminal prohormone of brain natriuretic peptide (NT-proBNP) will be obtained via blood draw. This will be assessed at approximately six months post-Barostim titration and compared with the NT-proBNP levels obtained during the pre-implantation phase. Change from baseline will be calculated.
Change in sleep score at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  The most recent 30-day average of sleep scores will be measured via study-provided Fitbit Inspire 3 fitness trackers. This sleep score is calculated by Fitbit as a proprietary algorithm to assess sleep quality based upon time asleep, time in sleep stages, movement during sleep, and sleeping heart rate, derived from measurements obtained by the fitness tracker. It is a score graded from 0-100, with 100 being the best score. This will be assessed at approximately six months post-Barostim titration and compared with the proportion of exercise days of the last 30-day period prior to the end of the pre-implantation phase. Change from baseline will be calculated.
Change in heart failure admissions at 6 months post-titration | Pre-implantation phase (baseline, approximately 0 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Participants' heart failure-related hospital admission counts will be obtained for the preceding six months at each time point. This will be calculated at approximately six months post-Barostim titration and compared with the same calculation of admissions at the time of study intake. Change from baseline will be calculated.

OTHER OUTCOMES:
Correlate estimated peak VO2 by smartwatch to peak VO2 obtained via cardiopulmonary exercise testing | Pre-implantation phase (baseline, approx. 2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Participants' cardio fitness score (estimated peak VO2) will be compared for correlation to peak VO2 measurements obtained from cardiopulmonary exercise testing (CPET). The most recent cardio fitness score will be measured via study-provided Fitbit Inspire 3 fitness trackers to correspond temporally with the date of the CPET study. Correlations will be assessed separately at each time point, i.e., approximately six months post-Barostim titration and during the pre-implantation phase. Correlations will also be assessed using data from both time points.
Change in estimated peak VO2 by smartwatch after implantation over time | Pre-implantation phase (baseline, 0-2 months) and post-implantation phase (approximately 0-9 months post-implantation) at regular intervals, e.g., monthly
  Participants' cardio fitness scores (estimated peak VO2) will be collected at regular intervals before and after implantation of the Barostim device. The cardio fitness scores will be measured via study-provided Fitbit Inspire 3 fitness trackers. These scores will be compared for trend over time.
Change in clinically significant echocardiography parameters at 6 months post-titration | Pre-implantation phase (baseline, 0-2 months) and post-titration phase (approximately 6 months after completion of device titration, i.e. approx. 7-9 months post-implantation).
  Echocardiography will be obtained at approximately six months post-Barostim titration and compared with echocardiography measured during the pre-implantation phase. Measurements such as left and right atrial size; left and right ventricular size and systolic function; and presence and degree of aortic, mitral, tricuspid, and pulmonic stenosis or regurgitation will be compared. Change from baseline will be calculated.
Time to completion of Barostim device titration | Implantation and titration phases, to complete approximately 3 months after device implantation.
  Each participant's time to device titration will be obtained and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Uriel, MD, Principal Investigator — Columbia University
Locations (7):
- United States (7):
  - University of California San Francisco Health, San Francisco, California
  - MedStar Health, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - Weill Cornell Medicine, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - Medical University of South Carolina Health, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data underlying the results reported in publications may be shared with qualified researchers upon reasonable request, following publication of the primary study results. Requests will be reviewed by the study investigators and, if approved, data will be shared under a data use agreement and in accordance with applicable institutional and regulatory requirements.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Zile MR, Lindenfeld J, Weaver FA, Zannad F, Galle E, Rogers T, Abraham WT. Baroreflex Activation Therapy in Patients With Heart Failure With Reduced Ejection Fraction. J Am Coll Cardiol. 2020 Jul 7;76(1):1-13. doi: 10.1016/j.jacc.2020.05.015. PMID 32616150
- [Background] Coats AJS, Abraham WT, Zile MR, Lindenfeld JA, Weaver FA, Fudim M, Bauersachs J, Duval S, Galle E, Zannad F. Baroreflex activation therapy with the Barostim device in patients with heart failure with reduced ejection fraction: a patient level meta-analysis of randomized controlled trials. Eur J Heart Fail. 2022 Sep;24(9):1665-1673. doi: 10.1002/ejhf.2573. Epub 2022 Jul 3. PMID 35713888
- See also: Summary of Safety and Effectiveness Data (SSED; FDA) — https://www.accessdata.fda.gov/cdrh_docs/pdf18/P180050b.pdf